CLINICAL TRIAL: NCT05359042
Title: Electronic Patient Reported Outcomes in Patients With Gastrointestinal Cancers at Risk for Unplanned ED Visits and Hospitalizations
Brief Title: Electronic Patient Reported Outcomes in Patients With Gastrointestinal Cancers
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Logistical constraints
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 214511; NCI-2022-02553 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2022-04-27; First posted 2022-05-03 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Gastrointestinal Cancers; Gastrointestinal Cancer Metastatic
Keywords: Patient Reported Outcomes; Hospitalizations; Emergency Department Visits
MeSH Terms: conditions — Gastrointestinal Neoplasms | interventions — Quality of Life

STUDY DESIGN:
Intervention Model Description: Patients will be randomized 2:1 to intervention arm or the standard of care arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ePRO Assessment Tool (Experimental): Participants will receive either a text message or an email inviting them to engage in the health chat. Participant assessments including HRQOL and user experience will be administered via the platform. Participants will also be able to participate in short, interactive patient education modules related to the infusion and side effect management.
  Interventions: Other: Electronic Patient Reported Outcomes platform; Other: Health Related Quality of Life Surveys
- Standard of Care (No Intervention): Participants in the standard of care arm will report symptoms via standard of care messaging through UCSF MyChart or telephone calls throughout the study period, and complete standard of care HRQoL surveys.

INTERVENTIONS:
Other: Electronic Patient Reported Outcomes platform — The ePRO tool is developed by a third-party vendor, Conversa, and engages the patient in a chat-based interaction to assess patient symptoms and provide educational material.
  Other Names: ePRO platform
  Arms: ePRO Assessment Tool
Other: Health Related Quality of Life Surveys — Surveys will be administered to participants
  Other Names: HRQoL
  Arms: ePRO Assessment Tool

SUMMARY:
This is a randomized trial of patients with gastrointestinal (GI) cancers treated at University of California, San Francisco (UCSF) who are starting a new line of systemic therapy to evaluate the feasibility of electronic patient reported outcome (ePRO) platform.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the feasibility of the ePRO platform by describing the proportion of participants who engage with the ePRO tool via virtual care chat at least once after enrollment.

II. To investigate the potential differences in health-related quality of life (HRQoL) by comparing the change in overall score of EuroQol five-dimensional Questionnaire (EQ-5D) index.

SECONDARY OBJECTIVES:

I. To evaluate the degree of engagement with virtual care chat as defined by the proportion of chat modules completed.

II. To measure the potential differences in health-related quality of life (HRQoL).

III. To describe the symptom experience of participants in the intervention arm.

IV. To evaluate the performance of clinical escalation rules and impact on clinic workflow and efficiency.

V. To prospectively validate a risk model predicting emergency department (ED) visits and admissions due to cancer treatment side effects.

EXPLORATORY OBJECTIVES:

I. To compare unplanned ED visits and hospitalizations between intervention arm and control arm.

II. To compare referral patterns to Symptom Management Clinic. III. To compare concordance between participant self-reported and provider assigned Eastern Cooperative Oncology Group (ECOG) Performance Status.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older
* Diagnosis of gastrointestinal cancers: esophageal, gastric, hepatocellular carcinoma, cholangiocarcinoma, pancreatic, neuroendocrine, small intestine, colorectal and anal cancers.
* Patients can have early stage or advanced cancer and will be starting treatment with new, standard of care infusion therapy regimen at UCSF.
* Ability to understand study procedures and to comply with them for the entire length of the study.
* No limit on prior lines of therapy.
* Access to smartphone, tablet, or computer with capability to use symptom tracking web site (must have mobile phone number or email address).
* Willing and able to provide written, signed informed consent in English.
* Ability of individual or legal guardian/representative to understand a written informed consent document, and the willingness to sign it.

Exclusion Criteria:

* Patients who have already started therapy prior to study enrollment.
* Patients who are receiving their treatment outside of UCSF.
* Participation in another clinical trial (therapeutic or non-therapeutic).
* Patients who are on therapy with oral oncolytics or combination therapy of oral oncolytics and infusional agents.
* Patients who are non-English speakers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-06-15 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who engaged with the ePRO tool | Up to 6 months
  The point estimation of proportion of patients who engaged with the ePRO tool via virtual care chat at least once after enrollment and its 95% binomial confidence interval (CI) will be obtained.
Change in overall score of EQ-5D | 6 months
  The EQ-5D is a standardized instrument for measuring generic health status. The health status is measured in terms of five dimensions (5D); mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The respondents self-rate their level of severity for each dimension by selecting one of the following responses: no problems (0), slight problems (1), mild problems (2), moderate problems (3), or severe problems (4) with a particular dimension. Lower scores indicate less issues/problems with that particular health dimension. Change in overall score of EQ-5D index between the intervention and usual of care arms between baseline and 6 months will be reported

SECONDARY OUTCOMES:
Proportion of chat modules completed | Up to 6 months
  To evaluate the degree of engagement with virtual care chat as defined by the proportion of chat modules completed per patient. Point estimation and 95% binomial CI will be obtained assuming normality assumption holds.
Proportion of chats in which PRO-CTCAE was offered were completed. | Up to 6 months
  To evaluate the degree of engagement with virtual care chat as defined by the proportion of chats in which PRO-CTCAE was offered were completed. Point estimation and 95% binomial CI will be obtained assuming normality assumption holds
Change in EQ-5D scores over time | Up to 6 months
  The EQ-5D is a standardized instrument for measuring generic health status. The health status is measured in terms of five dimensions (5D); mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The respondents self-rate their level of severity for each dimension by selecting one of the following responses: no problems (0), slight problems (1), mild problems (2), moderate problems (3), or severe problems (4) with a particular dimension. Lower scores indicate less issues/problems with that particular health dimension. Change in overall score of EQ-5D index between the intervention and usual of care arms between baseline, every 3 months, and at the completion of the study will be examined using a linear mixed model.
Number of patient-reported symptoms | Up to 6 months
  Number of patient-reported symptoms over the 6-month study period will be reported by frequency of symptom.
Number of patient-reported symptoms that were severe and were escalated | Up to 6 months
  Number of patient-reported symptoms that were categorized as severe and escalated will be reported by frequency of symptom.
Mean change in pain score over time. | Up to 6 months
  The pain score will be obtained using a standard pain index with values ranging from 0= No Pain to 10= Worst pain as reported by patients. Higher scores indicate a greater degree of patient reported pain. The change in pain scores will be evaluated using a linear mixed model.
Number of phone calls and secure messages | Up to 6 months
  The overall volume of phone calls and secure messages between each patient and the clinical team will be reported.
Predictive value of ED Visit and/or hospital admission | Up to 6 months
  To prospectively validate a risk model predicting ED visits and admissions due to treatment side effects via Model area under the receiver operating characteristic (AUROC). Accuracy of a previously developed model will be prospectively assessed during the course of this study. The model currently generates an assessment of risk that a patient will have an Chemotherapy Measure (OP-35) qualifying event in the 30-day period following an infusional therapy administration. An OP-35 event is defined as: One or more inpatient admissions for anemia, dehydration, diarrhea, emesis, fever, nausea, neutropenia, pain, pneumonia, or sepsis within 30 days of chemotherapy treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Wesley A Kidder, MD, Principal Investigator — University of California, San Francisco

IPD SHARING:
Plan to Share IPD: No